CLINICAL TRIAL: NCT01204372
Title: Phase II Trial Evaluating the Combination of Gemcitabine, Trastuzumab and Erlotinib as First-line Chemotherapy in Patients With Metastatic Pancreatic Adenocarcinoma
Brief Title: Trial Evaluating Combined Chemotherapy in Patients With Metastatic Pancreatic Adenocarcinoma
Acronym: GATE 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GATE 1; 2009-016875-30 (EudraCT Number)
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: Metastatic pancreatic adenocarcinoma; First-line chemotherapy; Combination chemotherapy; Targeted agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Gemcitabine - Trastuzumab - Erlotinib
  Interventions: Drug: Gemcitabine - Trastuzumab - Erlotinib

INTERVENTIONS:
Drug: Gemcitabine - Trastuzumab - Erlotinib — Treatment will be administered until disease progression, patient's refusal, unacceptable toxicity or investigator's decision.
  * Gemcitabine: IV 1000 mg/m2 on D1, D8, D15, D22, D29, D36 and D43 followed by one week of rest. Subsequently on D1, D8 and D15 followed by one week of rest.
  * Trastuzumab: IV once a week; 4 mg/kg over 90 min. at D1, and 2 mg/kg over 30 min. for the subsequent infusions.
  * Erlotinib: oral route 100 mg/day from C1D1.

SUMMARY:
GATE 1 is an open-label, non-comparative, multicentric study evaluating the efficacy and tolerance of the combined use of Gemcitabine, Trastuzumab and Erlotinib as a first-line chemotherapy in metastatic pancreatic cancer patients.

The patients will be treated intravenously with Gemcitabine at a dose of 1000 mg/m2 for 30 min. For the first eight weeks, Gemcitabine will be administered once weekly for 7 weeks followed by one week of rest. Subsequently, Gemcitabine will be administered once weekly for three weeks followed by one week of rest.

Trastuzumab will be administered once a week at a dose of 4 mg/kg over 90 min. at D1 and then at 2 mg/kg over 30 min. for the subsequent infusions.

Erlotinib will be administered orally at a dose of 100 mg/day from C1D1.

The patients will be subjected to research for the EGFR, HER2 and KRAS status.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic pancreatic adenocarcinoma confirmed by histology
* Tumor sample available
* Measurable lesion according to RECIST criteria
* Performance status ≥ 1
* Life expectancy > 3 months
* Hematology: Hb ≥ 9g/dL, neutrophils ≥ 1,500/mm3, platelets ≥ 100,000/mm3
* Renal function: creatinine ≤ 1.5 x ULN
* Hepatic function: total bilirubin ≤ 2.5 x ULN, transaminases ≤ 5 x ULN
* Left ventricular ejection fraction (LVEF) ≥ 50%
* At least a 6-month delay between the end of any previous gemcitabine-based chemotherapy and diagnosis of metastases
* Social security
* Informed consent obtained prior to inclusion.

Exclusion Criteria:

* Non metastatic advanced local disease
* Presence of cerebral metastases or symptomatic leptomeningeal carcinomatosis
* Others cancers except BBC and cervical cancer receiving curative treatment
* No previous treatment by Erlotinib or Trastuzumab
* Known severe hypersensitivity to Erlotinib, Trastuzumab, murine proteins or Gemcitabine
* Presence of significant co-morbidities
* Concomitant treatment with other experimental products or other anticancer therapies
* Breastfeeding or pregnant female, or patient of reproductive age not using adequate contraception
* Legal incapacity or limited legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Disease control rate according to RECIST criteria of the Gemcitabine, Trastuzumab and Erlotinib combination. | Every 8 weeks and at the treatment completion
  The tumor evaluation will be based on:
  * Clinical examination
  * TAP CT-scan or MRI
  * Tumor marker dosage (CEA and CA 19-9)

SECONDARY OUTCOMES:
Progression free survival | Every 8 weeks and at the treatment completion
  The tumor evaluation will be based on:
  * Clinical examination
  * TAP CT-scan or MRI
  * Tumor marker dosage
Overall survival | Every 8 weeks and at treatment completion

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Val d'Aurelle, Montpellier, France

REFERENCES:
- [Derived] Assenat E, Mineur L, Mollevi C, Lopez-Crapez E, Lombard-Bohas C, Samalin E, Portales F, Walter T, de Forges H, Dupuy M, Boissiere-Michot F, Ho-Pun-Cheung A, Ychou M, Mazard T. Phase II study evaluating the association of gemcitabine, trastuzumab and erlotinib as first-line treatment in patients with metastatic pancreatic adenocarcinoma (GATE 1). Int J Cancer. 2021 Feb 1;148(3):682-691. doi: 10.1002/ijc.33225. Epub 2020 Sep 2. PMID 33405269